CLINICAL TRIAL: NCT04233424
Title: D-PLEX 311- Phase III, Prospective, Multinational, Multicenter, Randomized, Controlled, Two-arm, Double Blind Study to Assess Efficacy and Safety of D-PLEX In Prevention of Post Abdominal Surgery Incisional Infection(SHIELD I)
Brief Title: D-PLEX 311: Safety and Efficacy of D-PLEX in the Prevention of Post Abdominal Surgery Incisional Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PolyPid Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D-PLEX 311
Record Dates: First submitted 2020-01-06; First posted 2020-01-18 (Actual); Results first posted 2025-06-22 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Surgical Site Infection; Colon Surgery; Abdominal Surgery; Post-Op Infection
Keywords: Surgical site infection; Abdominal surgery; Colon and small bowl surgery
MeSH Terms: conditions — Surgical Wound Infection | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Males and females, >18 years old, undergoing scheduled abdominal colon surgery involving resection and anastomosis or a stoma, who meet the inclusion criteria and none of the exclusion criteria and provide signed informed consent will be enrolled in the study.
  The final number of subjects will be determined following a comparative interim analysis for an early efficacy or futility stop or unblinded sample size re-estimation: when about 750 subjects will complete their 30 days (1 month) follow-up and evaluated for primary endpoint.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind clinical trial. The sponsor, the subjects, outcomes assessor and all staff involved in the collection and recording of the clinical and laboratory data, based on which the independent adjudication committee will perform their assessment, will be blind to treatment assignment. In addition, all aspects of data management and clean-up will be done in blinded datasets.
  The study site personnel, who perform the index surgery (Operation room staff), will be trained not to disclose the treatment arm to the blinded Investigator, to the subject, his/her family, to other health care providers not present during the surgery or to the study Sponsor representatives. Wound assessment throughout the study follow-up visits will be done by a blinded Investigator, that will not be involved in the surgery. An emergency card containing the Study Name, NIH number, Center Name/number, PI's name and contact details will be provided to the subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- D-PLEX+SoC (Experimental): D-PLEX is provided to suitable and willing study subjects as an adjunct to the SoC treatment
  Interventions: Drug: D-PLEX; Drug: Standard of Care (SoC)
- Standard of care (Other): The SoC for prophylactic antibiotic treatment is based on international guidelines
  Interventions: Drug: Standard of Care (SoC)

INTERVENTIONS:
Drug: D-PLEX — D-PLEX is a new formulation of extended release of Doxycycline. Each 5g D-PLEX vial contains 54.6mg Doxycycline free base (1.09%), which is equivalent to 63mg Doxycycline hyclate (1.26%). D-PLEX is supplied as a sterile powder to be reconstituted to paste in the operating room, using standard aseptic techniques and is intended for single administration. The non-active components of the extended release antibiotic formulation are β Tri-Calcium polymer and a lipid matrix. All formulation components are biodegradable.
  Arms: D-PLEX+SoC
Drug: Standard of Care (SoC) — prophylactic, pre-operation per institution guidelines

SUMMARY:
Phase III, Prospective, Multinational, Multicenter, Randomized, Controlled, Two-arm, Double Blind Study to assess Efficacy and Safety of D-PLEX Administered Concomitantly with the Standard of Care (SoC), compared to a SoC treated control arm, in prevention of post abdominal surgery incisional infection.

DETAILED DESCRIPTION:
D-PLEX is a new formulation of extended controlled release of Doxycycline in the applied area for about 30 days. This study is aimed to assess the safety and efficacy of D-PLEX in prevention of post abdominal surgery incisional infection.

The study population includes male and female, 18 years old and above at screening, undergoing an elective colorectal surgery involving resection, with or without a stoma, that includes at least 1 incision that is > 10 cm (target incision). Eligible and willing subjects will be randomly allocated into 2 blinded study arms D-PLEX with SOC or SOC alone.

D-PLEX will be applied during the surgery at the final stage of incision closure. All patients will be followed up for additional 5 visits over 2 months, for safety and incisional wound assessment. This will include blood tests for hematology and chemistry well as physicians assessment of the incisional wound.

The final number of subjects will be determined following a comparative interim analysis for an early efficacy or futility stop or unblinded sample size re-estimation: when about 750 subjects will complete their 30 days (1 month) follow-up and evaluated for primary endpoint

ELIGIBILITY:
INCLUSION CRITERIA:

1. Subjects undergoing an elective colorectal surgery involving resection, with or without a stoma formation, that includes at least 1 abdominal incision that is > 10cm (target incision).
2. Subjects are preoperative hemodynamically stable
3. Male or non-pregnant female.
4. Female of child-bearing potential should have a negative pregnancy test prior to index procedure.
5. Subjects' age 18 years old and above at screening.
6. Subjects who sign the written Informed Consent Form.
7. Subjects who are willing and able to participate and meet all study requirements.
8. Survival expectancy of at least 60 days post randomization

EXCLUSION CRITERIA

1. Subjects with suspected/diagnosed intestinal perforation, intra-abdominal abscess, or any emergency/urgent colorectal surgery with acute intestinal obstruction (ex. toxic colitis, ileus/sub-ileus, megacolon, diverticulitis, volvulus, ect.)
2. Subjects who underwent an intra-abdominal surgery within the last 6 months prior to randomization.
3. Subjects with any preoperative active infection or who are receiving any antibiotic therapy in the past 1 week prior to randomization, excluding pre-operative prophylaxis.
4. Subjects undergoing concomitant major procedures in addition to the abdominal surgery, including concomitant repair of ventral hernia. Salpingo-oophorectomy and cholecystectomy are allowed.
5. Subjects who received any anti-cancer treatment within the last 4 weeks of surgery.
6. Subjects who received radiation for colorectal cancer to the abdomen area, prior to the planned abdominal surgery.
7. Subjects who received oral or IV Doxycycline or Tetracycline family antibiotics during the past 4 weeks prior to randomization.
8. Subjects with known allergy to Doxycycline and/or to the tetracycline family of drugs or to the D-PLEX's excipients.
9. Subjects with known allergies to more than 3 substances (an allergy questionnaire will be completed during the screening process).
10. Subjects with history of severe allergic reaction to any substance, having required treatment with intravenous steroids/intramuscular epinephrine, or who in the opinion of the PI is at high risk of developing severe allergic reactions.
11. Subjects with End Stage Renal Disease (ESRD/ CKD stage 5).
12. Subjects with severe hepatic impairment.
13. Subjects with chronic urticaria.
14. Subjects diagnosed with CVA within the past 6 months prior to randomization.
15. Subjects who underwent any abdominal surgery and current planned index surgery involves re-opening the scar of a prior abdominal surgery performed within the last 3 years.
16. Any subject with an active malignancy, other than resectable non-metastatic colorectal cancer, that is the reason for the index surgery, or carcinoma in situ (or other cancer "in situ = Stage 0"), or squamous cell carcinoma of the skin, or basal cell carcinoma of the skin, or a malignancy that has not been in complete clinical remission and without maintenance chemo or immunotherapy for at least 3 years.
17. Subjects with other concurrent severe and/or uncontrolled medical conditions.
18. Psychiatric or any other disorder that compromises ability to provide informed consent for participation in this study.
19. Chronic alcoholic or drug abuse subjects.
20. Pregnant or breast-feeding women or women of child-bearing age who refuse or are prohibited of using an effective contraceptive method of birth control throughout study participation, including the safety follow-up period.
21. Subjects who received any investigational drug within 30 days or 5 half-lives prior to randomization to the study (whichever is longer) and through the study.
22. Subjects participating in any other interventional study.
23. Subjects, who in the opinion of Investigator, are not eligible to participate in the study and/or to comply with the protocol requirements (e.g. due to a cognitive or medical condition).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 977 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shmuel Sharoni, MD, Study Director — PolyPid Ltd.
Locations (62):
- United States (5):
  - Shoals Medical Trials, Sheffield, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Paradigm Clinical Research Center, Redding, California
  - Tufts Medical Center, Boston, Massachusetts
  - Summit Medical Group, Bend, Oregon
- Bulgaria (12):
  - "Multiprofile Hospital for Active Treatment - Blagoevgrad" AD, Blagoevgrad
  - "Multiprofile Hospital for Active Treatment "Sveti Ivan Rilski - 2003" OOD, Dupnitsa
  - "Multiprofile Hospital for Active Treatment - Haskovo" AD, Haskovo
  - "Multiprofile Hospital for Active Treatment - Uni Hospital" OOD, Panagyurishte
  - "MHAT Sveta Caridad" EAD, Plovdiv
  - University First Multiprofile Hospital for Active Treatment - Sofia Sv. Yoan Krastitel EAD, Sofia
  - "IV Multiprofile Hospital for Active Treatment - Sofia" EAD, Sofia
  - "University Multiprofile Hospital for Active Treatment and Emergency Medicine N. I. Pirogov" EAD, Sofia
  - "Multiprofile Regional Hospital for Active Treatment "Dr. St. Cherkezov"" AD, Veliko Tarnovo
  - Complex Oncology Center - Vratsa - EOOD, Vratsa
  - Department - Surgery, "Multiprofile Hospital for Active Treatment - Hristo Botev" AD, Vratsa
  - "Multiprofile Hospital for Active Treatment "Sveti Panteleymon"-Yambol AD, Yambol
- Croatia (4):
  - KBC Rijeka, Rijeka
  - General Hospital Zadar, Zadar
  - KBC Sestre milosrdnice Klinika za tumore, Zagreb
  - University Hospital Centre Zagreb (KBC Rebro), Zagreb
- Czechia (4):
  - Fakultni Nemocnice Brno Chirurgicka klinika, Brno
  - Krajska nemocnice Liberec, a. s., Liberec
  - Fakultni nemocnice Kralovske Vinohrady Chirurgicka klinika, Prague
  - Nemocnice Na Bulovce, Prague
- Hungary (8):
  - Bajai Szent Rókus Kórház, Sebészeti Osztály, Baja, Bács-Kiskun Megye
  - Semmelweis Egyetem Altalanos Orvostudomanyi Kar, Sebeszeti es Intervencios Gasztroenterologiai, Budapest
  - Békés-Megyei Központi Kórház, I. Sebészeti Osztály, Gyula
  - Csongrad-Csanad Megyei Egeszsegugyi Ellato Kozpont Hodmezovasarhely - Mako, Sebeszeti Osztaly, Hódmezővásárhely
  - Somogy Megyei Kaposi Mór Oktató Kórház, Sebészeti Osztály, Kaposvár
  - Orosházi Kórház, Invazív Mátrix Sebészet, Orosháza
  - Pécsi Tudományegyetem, Klinikai Központ, Sebészeti Klinika, Pécs
  - Fejér Megyei Szent György Egyetemi Oktató Kórház, Sebészeti Osztály, Székesfehérvár
- Israel (7):
  - The Chaim Sheba Medical Center, Ramat Gan, Derech Sheba 2
  - Galilee Medical Center, Nahariya, Nahariya-Cabri
  - Kaplan Medical Center, Rehovot, Pasternak
  - Rabin Medical Center, Petah Tikva
  - Assuta Medical center, Tel Aviv
  - Sourasky Medical Center, Tel Aviv
  - Shamir (Assaf-Harofeh) Medical Center, Zrifin
- Moldova (5):
  - IMSP Institute of Emergency Medicine, Chisinau
  - IMSP Clinical Republican Hospital "Timofei Mosneaga", Chisinau
  - IMSP Institute of Oncology, Chisinau
  - IMSP Municipal Clinical Hospital "Sfanta Treime", Chisinau
  - PMSI Municipal Clinical Hospital No. 1 "Gheorghe Paladi" Department of General Surgery, Chisinau
- Poland (4):
  - Oddzial Kliniczny Chirurgii Onkologicznej, Bydgoszczy, Bydgoszcz
  - Szpital Specjalistyczny im. Zeromskiego,Oddzial Chirurgii Ogolnej Onkologicznej i Maloinwazyjnej, Krakow
  - Szpital Skawina Sp. z o.o., im. Stanley Dudricka, Skawina
  - Oddzial Chirurgii Ogolnej i Onkologicznej, Szpital Uniwersytecki im.Karola Marcinkowskiego, Zielona Góra
- Romania (10):
  - "Sf. Constantin" Hospital, Brasov
  - Emergency University Hospital Elias, Clinical Department of General Surgery, Bucharest
  - Coltea Clinical Hospital, Department of General Surgery, Bucharest
  - "Prof. Dr. Octavian Fodor", Cluj-Napoca
  - Medical Center Dr.Ianosi, Department of Surgery, Craiova
  - County Emergency Clinical Hospital Craiova, Department of General Surgery III, Craiova
  - County Emergency Clinical Hospital Craiova, Department of General Surgery II, Craiova
  - County Emergency Clinical Hospital Craiova, Department of General Surgery I, Craiova
  - Spitalul Clinic Judetean de Urgentã Targu-Mures, Craiova
  - County Emergency Clinical Hospital Timisoara "Pius Brînzeu", Timișoara
- Slovakia (3):
  - Vseobecna Nemocnica s Poliklinikou Lucenec Chirurgicke Oddelenie, Lučenec
  - FNsP J.A. Reimana Presov Oddelenie chirurgie, Prešov
  - Fakultna nemocnica s poliklinikou Zilina Oddelenie chirurgie, Žilina

RESULTS

PARTICIPANT FLOW:
Groups:
- D-PLEX+SoC: D-PLEX is provided to suitable and willing study subjects as an adjunct to the SoC treatment
  D-PLEX: D-PLEX is a new formulation of extended release of Doxycycline.
Period: Overall Study
Arm/Group | D-PLEX+SoC | Standard of Care
Started | 488 | 489
Number of Subjects in the ITT Population | 485 | 489
Actual number of subjects treated in each treatment group | 478 | 498
Completed | 464 | 458
Not Completed | 24 | 31
Not completed — Death | 15 | 16
Not completed — Withdrawal by Subject | 2 | 8
Not completed — Physician Decision | 1 | 3
Not completed — Protocol Violation | 3 | 1
Not completed — Lost to Follow-up | 1 | 3
Not completed — subject refuse to visit site | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to treat population (ITT) excluded 3 subjects which surgery plan was changed before surgery and abdominal incision was not performed.
Groups:
- Total: Total of all reporting groups
Arm/Group | D-PLEX+SoC | Standard of Care | Total
Number analyzed (Participants) | 485 | 489 | 974
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (12.75) | 63.7 (13.27) | 64.2 (13.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197 | 198 | 395
  Male | 288 | 291 | 579
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 483 | 486 | 969
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Romania | 82 | 86 | 168
  Hungary | 84 | 76 | 160
  United States | 18 | 19 | 37
  Czechia | 64 | 67 | 131
  Moldova | 84 | 93 | 177
  Israel | 67 | 71 | 138
  Bulgaria | 47 | 45 | 92
  Croatia | 26 | 14 | 40
  Poland | 8 | 9 | 17
  Slovakia | 5 | 9 | 14
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.80 (4.54) | 27.11 (4.65) | 26.96 (4.60)

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Anti-infective Efficacy of D-PLEX Over a Period of 30 Days Post Operation, by Preventing Surgical Site Infection (SSI), Defined as Superficial and Deep Infection, in the Target Incision(s), Compared to the SoC Treated Control.
Description: Infection rate as measured by the proportion of subjects with at least one abdominal incisional infection event, as determined by a blinded and independent adjudication committee, within 30 days post-abdominal surgery. [Abdominal incisional infection is composed of Deep Incisional Surgical Site Infection (DSSI) and Superficial Incisional Surgical Site Infection (SSSI)]. The blinded and independent adjudication committee review will include all index surgery incisions, regardless of any re-intervention at the target site, for the determination of infection status. The committee will also assess re-interventions at the primary incision site through the abdominal incision (target) for the determination of re-intervention due to suspected SSI or due to poor wound healing, including wound dehiscence. Such events, as well as all-cause mortality within 30 days post-index surgery will be analyzed as treatment failure.
Time Frame: By day 30 post surgery
Population: Intent to treat population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | D-PLEX+SoC | Standard of Care
Number analyzed (Participants) | 485 | 489
percentage of participants | 9.3 [6.8 to 12.2] | 12.1 [9.3 to 15.3]
Statistical Analysis 1: Comparison: D-PLEX+SoC vs Standard of Care; Test type: Superiority; p = 0.152, Cochran-Mantel-Haenszel; Risk Ratio (RR) = -2.8, 95% CI 2-sided [-6.7 to 1.0]

2. Secondary Outcome: Assessment of Infection Rate in Patient Undergoing Abdominal Colon Surgery
Description: infection rate as measured by the proportion of subjects with at least one abdominal incisional infection event, as determined by a blinded and independent adjudication committee, within 30 days post abdominal surgery. [abdominal incisional infection is composed of Deep Incisional Surgical Site Infection (DSSI) and Superficial Incisional Surgical Site Infection (SSSI)].
Time Frame: 30 days post-surgery
Population: Intent to treat population
Measure: Number (95% Confidence Interval); unit: Percentage of the participants
Arm/Group | D-PLEX+SoC | Standard of Care
Number analyzed (Participants) | 485 | 489
Percentage of the participants | 6.2 [4.2 to 8.8] | 6.9 [4.7 to 9.5]
Statistical Analysis 1: Comparison: D-PLEX+SoC vs Standard of Care; Test type: Superiority; p = 0.6219, Cochran-Mantel-Haenszel; Risk Ratio (RR) = -0.8, 95% CI 2-sided [-3.9 to 2.3]

3. Other Pre Specified Outcome: All-cause Mortality
Description: All-cause mortality within 30 days post index surgery will be analysed as treatment failure.
Time Frame: 30 day post surgery
Population: All-cause mortality is calculated out of the ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | D-PLEX+SoC | Standard of Care
Number analyzed (Participants) | 485 | 489
percentage of participants | 2.3 [1.3 to 4.1] | 3.1 [1.9 to 5.1]
Statistical Analysis 1: Comparison: D-PLEX+SoC vs Standard of Care; Test type: Superiority; p = 0.4373, Kaplan-Meier Analysis; Risk Ratio (RR) = -0.8, 95% CI 2-sided [-2.8 to 1.2]

ADVERSE EVENTS:
Time Frame: 60 days
Description: Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. "Lack of efficacy" or "failure of expected pharmacology action" per se will not be reported as an AE or SAE. However, the signs and symptoms and/or clinical sequelae resulting from lack of efficacy will be reported if they fulfil the definition of an AE or SAE.
Arm/Group | D-PLEX+SoC | Standard of Care
All-Cause Mortality (participants affected / at risk) | 16/485 | 17/489
Serious Adverse Events (participants affected / at risk) | 69/478 | 98/498
Other Adverse Events (participants affected / at risk) | 381/478 | 398/498
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-PLEX+SoC (N=478) | Standard of Care (N=498)
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anastomotic leak (Injury, poisoning and procedural complications) | 8 (8) | 19 (19)
Cardiac failure (Cardiac disorders) | 2 (2) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 6 (6)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 2 (2)
Cardiopulmonary failure (Cardiac disorders) | 2 (2) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2) | 5 (5)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 4 (4)
Gastrointestinal necrosis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Intestinal fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal ischemia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 3 (3)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Hepatorenal failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 8 (8) | 6 (6)
Peritonitis (Infections and infestations) | 4 (4) | 5 (5)
Pneumonia (Infections and infestations) | 4 (4) | 5 (5)
Abdominal abscess (Infections and infestations) | 4 (4) | 4 (4)
COVID-19 (Infections and infestations) | 6 (6) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 4 (4)
Septic shock (Infections and infestations) | 1 (1) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pelvic abscess (Infections and infestations) | 2 (2) | 0 (0)
Device related bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Endotoxic shock (Infections and infestations) | 1 (1) | 0 (0)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0)
Mediastinitis (Infections and infestations) | 0 (0) | 1 (1)
Necrotizing fasciitis (Infections and infestations) | 1 (1) | 0 (0)
Medical device site infection (Infections and infestations) | 0 (0) | 1 (1)
Pelvic infection (Infections and infestations) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Acinetobacter Baumanni (Infections and infestations) | 0 (0) | 1 (1)
Purulent discharge (Infections and infestations) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Stoma site infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Anastomotic complication (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Wound evisceration (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Anastomotic fistula (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Anastomotic hemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Abdominal wall wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Carcinogenicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ureteric injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Ischemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Orchitis noninfective (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic fluid collection (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemodynamic instability (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-PLEX+SoC (N=478) | Standard of Care (N=498)
Anaemia (Blood and lymphatic system disorders) | 12 (12) | 15 (15)
Tachycardia (Cardiac disorders) | 13 (15) | 7 (7)
Nausea (Gastrointestinal disorders) | 41 (42) | 52 (56)
Vomiting (Gastrointestinal disorders) | 29 (30) | 21 (23)
Abdominal Pain (Gastrointestinal disorders) | 21 (21) | 17 (17)
Diarrhea (Gastrointestinal disorders) | 19 (20) | 18 (18)
Abdominal Distension (Gastrointestinal disorders) | 6 (6) | 11 (11)
Constipation (Gastrointestinal disorders) | 6 (6) | 11 (12)
Ileus (Gastrointestinal disorders) | 7 (7) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 4 (4)
Abdominal Pain Upper (Gastrointestinal disorders) | 5 (5) | 3 (3)
Small Intestinal Obstruction (Gastrointestinal disorders) | 4 (4) | 6 (6)
Haematochezia (Gastrointestinal disorders) | 3 (3) | 5 (5)
Pain (General disorders) | 83 (83) | 85 (89)
Tenderness (General disorders) | 63 (63) | 64 (66)
Feeling Hot (General disorders) | 33 (33) | 33 (33)
Pyrexia (General disorders) | 16 (18) | 23 (23)
Swelling (General disorders) | 16 (16) | 23 (23)
Asthenia (General disorders) | 5 (5) | 11 (11)
Impaired Healing (General disorders) | 7 (7) | 1 (1)
Oedema Peripheral (General disorders) | 2 (2) | 6 (6)
Secretion Discharge (General disorders) | 5 (5) | 2 (2)
Postoperative Wound Infection (Infections and infestations) | 43 (45) | 52 (56)
Urinary Tract Infection (Infections and infestations) | 8 (8) | 16 (16)
COVID-19 (Infections and infestations) | 9 (10) | 13 (13)
Pneumonia (Infections and infestations) | 9 (9) | 9 (9)
Incision Site Pain (Injury, poisoning and procedural complications) | 111 (158) | 118 (167)
Procedural Pain (Injury, poisoning and procedural complications) | 83 (87) | 87 (91)
Incision Site Erythema (Injury, poisoning and procedural complications) | 52 (52) | 52 (53)
Incision Site Discharge (Injury, poisoning and procedural complications) | 53 (54) | 37 (37)
Incision Site Swelling (Injury, poisoning and procedural complications) | 25 (25) | 23 (23)
Anastomotic Leak (Injury, poisoning and procedural complications) | 11 (11) | 23 (23)
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 8 (8) | 5 (5)
Incision Site Haematoma (Injury, poisoning and procedural complications) | 7 (7) | 4 (4)
Wound dehiscence (Injury, poisoning and procedural complications) | 6 (6) | 5 (5)
Anastomotic Complication (Injury, poisoning and procedural complications) | 6 (6) | 3 (3)
Incision Site Haemorrhage (Infections and infestations) | 3 (3) | 5 (6)
Oxygen Saturation Decreased (Investigations) | 13 (13) | 16 (17)
Haemoglobin Decreased (Investigations) | 8 (8) | 11 (11)
C-reactive Protein Increased (Investigations) | 7 (7) | 7 (7)
Blood Albumin Decreased (Investigations) | 8 (8) | 4 (4)
SARS-CoV-2 Test Positive (Investigations) | 2 (2) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 11 (11) | 11 (11)
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 (7) | 4 (5)
Dizziness (Nervous system disorders) | 5 (5) | 2 (2)
Oliguria (Renal and urinary disorders) | 4 (4) | 5 (5)
Urinary Retention (Renal and urinary disorders) | 5 (5) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)
Hypertension (Vascular disorders) | 11 (11) | 7 (8)
Hypotension (Vascular disorders) | 7 (7) | 6 (6)
Haematoma (Vascular disorders) | 5 (5) | 1 (1)
Peritonitis (Infections and infestations) | 6 (6) | 9 (9)
Metastases to Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 8 (8)
Headache (Nervous system disorders) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/24/NCT04233424/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/24/NCT04233424/SAP_001.pdf